CLINICAL TRIAL: NCT04575298
Title: To Evaluate the Acceptability, Gastrointesinal Tolerance and Compliance of a Hypoallergenic Powdered Amino Acid Infant Formula with HMOs for the Dietary Management of Cows' Milk Allergy (CMA) and Multiple Food Allergies.
Brief Title: Acceptability and Tolerance Study of an Amino Acid Formula with HMOs
Status: Terminated | Type: Observational
Why Stopped: Difficulty to recruit patients due to pandemic
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: Alfamino with HMOs
Record Dates: First submitted 2020-03-06; First posted 2020-10-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Infant Development

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Dietary Supplement: Acceptability, tolerance study for an infant formula with human milk oligosaccharides — Prospective study

SUMMARY:
To evaluate the acceptability (including gastrointestinal tolerance and compliance) of a hypoallergenic amino acid infant formula with HMOs for the dietary management of cows' milk allergy in infants less than 12 months of age.

DETAILED DESCRIPTION:
This is an acceptability study to evaluate the gastrointestinal tolerance and compliance over a 7-day period, of Amino acid formula with HMOs, which is a hypoallergenic amino acid for infant formula for the dietary management of cows' milk allergy.

The acceptability data from a minimum of 15 participants will be collected in order to submit an application to the Advisory Committee on Borderline Substances (ACBS) and the HSE for the Ireland to be reimbursed under the GMS and community drug schemes

ELIGIBILITY:
Inclusion Criteria:

Patients well established and stable on Alfamino (or another amino acid formula dependent on feasibility of reaching required numbers) for the dietary management of presumed CMA (no gastrointestinal intolerances on current formula).

Full term infants less than 12 months of age where the amino acid formula is still the sole source of nutrition. Full term infants less than 12 months of age where the amino acid formula is required for 1 week to measure GI tolerance and 1 week of exclusive HMO amino acid formula intake. Thereafter formula intake data will be collected for the remaining 3 weeks and the child can be weaned at this stage.

iWillingly given, written, informed consent from patient or parent/guardian.

Exclusion Criteria:

Partially or fully Breastfed infants. Inability to comply with the study protocol, in the opinion of the investigator.

Previously not tolerated Alfamino without HMOs. More than 12 months old Need an amino acid formula as supplementary use Patients with significant renal or hepatic impairment Change in current medication or use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the investigator e.g. thickener, PPIs etc (must be recorded in patient case record file).

Participation in another interventional study within 2 weeks of this study. Introduction of complementary feeding during the study period Caregiver unable to read and write in English (will need to complete 7 1 monthdays of forms at home).

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | Day 7 from baseline
  Questionnaire to assess GI symptoms
Acceptability | Over a 28 days period recorded on a feeding chart
  Daily diary measuring volume of formula suggested versus actual formula taken

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Kakleas, Principal Investigator — Paediatric allergy consultant
Locations (1):
- Children's Research Team, Leicester, United Kingdom